CLINICAL TRIAL: NCT02725697
Title: Treatment of Acute and Chronic Complaints Following Sports Injuries With Traditional Chinese Medicine (TCM) by Therapists in Switzerland - a Prospective Observational Study
Brief Title: Treatment of Complaints Following Sports Injuries With Traditional Chinese Medicine
Status: Terminated | Type: Observational
Why Stopped: too few participans available
Sponsor: Sabine Klein (Other)
Responsible Party: Sponsor-Investigator, Sabine Klein, Head of Research Working Group, Swiss Professional Organization for Traditional Chinese Medicine
Organization: Swiss Professional Organization for Traditional Chinese Medicine (Other)
Other Study IDs: SBO-TCM 001
Record Dates: First submitted 2016-03-20; First posted 2016-04-01 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TCM treatment: TCM treatment (e.g. acupuncture, Tuina massage, Chinese herbal medicine, moxibustion, electroacupuncture, ear acupuncture)
  Interventions: Other: TCM treatment

INTERVENTIONS:
Other: TCM treatment

SUMMARY:
The purpose of this observational study is to investigate the treatment of complaints following sports injuries with Traditional Chinese Medicine by therapists in Switzerland.

DETAILED DESCRIPTION:
In Switzerland, still very little is known about the treatment with TCM (acupuncture, Chinese medicinal therapy, Tuina massage, nutrition, qigong) under everyday conditions. The importance of non-medical therapists in the healthcare system is rarely investigated. It is likely that patients with chronic injuries use several therapies (including conventional medicine) in a pragmatic way. They may apply TCM either due to primary preference or because other forms of therapy fail to produce satisfactory results.

There is evidence from randomized controlled trials and systematic reviews that acupuncture can be effective in the treatment of acute and chronic back pain, chronic shoulder pain and ankle sprains.

Randomized controlled trials usually investigate a single TCM method, in which therapists or physicians are limited in the selection of acupuncture points or herbal formulas. This does not reflect the complex practice, where several TCM methods and auxiliary techniques are combined.

The investigators aim to investigate in a prospective observational study how complaints following sports injuries are treated by non-medical TCM therapists in Switzerland under everyday conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* minimum of 3 hours sports per week
* complaints following sports injury
* first TCM treatment for this complaint

Exclusion Criteria:

* rheumatic disease
* arthrosis
* previous TCM treatment for this complaint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking TCM treatment due to complaints following sports injuries.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
change in minimal and maximal pain | first treatment, last treatment (max. 3 months)
  visual analogue scale (0-10)
change in limitation during sports | first treatment, last treatment (max. 3 months)
  visual analogue scale (0-10)

SECONDARY OUTCOMES:
medication intake | first treatment, last treatment (max. 3 months)
patient satisfaction with therapy | 6 months
  6 point Likert scale
number of therapeutic sessions | 3 months
TCM methods applied | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabine D Klein, PhD, Principal Investigator — Swiss Professional Organization for Traditional Chinese Medicine
Locations (3):
- Switzerland (3):
  - Poliklinik für Chinesische Medizin, Horgen, Canton of Zurich
  - Praxis für TCM, Zurich, Canton of Zurich
  - proSANUS, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein SD, Frei-Erb M, Wolf U. Usage of complementary medicine across Switzerland: results of the Swiss Health Survey 2007. Swiss Med Wkly. 2012 Aug 15;142:w13666. doi: 10.4414/smw.2012.13666. eCollection 2012. PMID 22895817
- [Background] Michlig M, Ausfeld-Hafter B, Busato A. Patient satisfaction with primary care: a comparison between conventional care and traditional Chinese medicine. Complement Ther Med. 2008 Dec;16(6):350-8. doi: 10.1016/j.ctim.2007.12.001. Epub 2008 Feb 4. PMID 19028336
- [Background] Lin ZP, Chen YH, Chia F, Wu HJ, Lan LW, Lin JG. Episodes of injuries and frequent usage of traditional Chinese medicine for Taiwanese elite wrestling athletes. Am J Chin Med. 2011;39(2):233-41. doi: 10.1142/S0192415X11008774. PMID 21476201
- [Background] Malone MA, Gloyer K. Complementary and alternative treatments in sports medicine. Prim Care. 2013 Dec;40(4):945-68, ix. doi: 10.1016/j.pop.2013.08.010. Epub 2013 Sep 26. PMID 24209727
- [Background] Park J, Hahn S, Park JY, Park HJ, Lee H. Acupuncture for ankle sprain: systematic review and meta-analysis. BMC Complement Altern Med. 2013 Mar 4;13:55. doi: 10.1186/1472-6882-13-55. PMID 23496981
- See also: Website of Swiss Professional Organization for Traditional Chinese Medicine — http://www.sbo-tcm.ch/